# Informed consent

#### Administrative information

Full study title Effects of dietary gluten on gastrointestinal symptoms in ulcerative colitis: a

randomised crossover trial.

Acronym Gluten-UC

Clinicaltrials.gov Identifier NCT06249763

Ethics Committee number S-20210174

The Danish Data Protecting

Agency Number 22/39335

Document date November 2<sup>nd</sup>, 2023

## **DET VIDENSKABSETISKE KOMITÉSYSTEM**

**(S4)** 

#### Informeret samtykke til deltagelse i et sundhedsvidenskabeligt forskningsprojekt.

Forskningsprojektets titel: Kostens betydning for patienter med inflammatorisk tarmsygdom; kan den glutenfri diæt lindre symptomerne og give mere energi i hverdagen?

### Erklæring fra forsøgspersonen:

Jeg har fået skriftlig og mundtlig information og jeg ved nok om formål, metode, fordele og ulemper til at sige ja til at deltage.

Jeg ved, at det er <u>frivilligt at deltage</u>, og at jeg altid kan trække mit samtykke tilbage uden at miste mine nuværende eller fremtidige rettigheder til behandling.

Jeg giver samtykke til, at deltage i forskningsprojektet og til, at mit biologiske materiale udtages med henblik på opbevaring i en forskningsbiobank. Jeg har fået en kopi af dette samtykkeark samt en kopi af den skriftlige information om projektet til eget brug.

| Forsøgspersonens navn: _ | |
|---|---|
| Dato: | Underskrift: |
| informeret. Vil du frabede | entlige helbredsoplysninger frem om dig i forskningsprojektet vil du blive<br>dig information om nye væsentlige helbredsoplysninger, som kommer frem i<br>du markere her: (sæt x) |
| Ønsker du at blive informe | ret om forskningsprojektets resultat samt eventuelle konsekvenser for dig?: |
| Ja (sæt x) Nej | (sæt x) |
| Efter min overbevisning er<br>deltagelse i forsøget. | fgiver information: rsonen har modtaget mundtlig og skriftlig information om forsøget. der givet tilstrækkelig information til, at der kan træffes beslutning om givet information: Laura Gregersen |
| Dato: | Underskrift: |
| · | omiteens Projekt-ID, EudraCT nr., versions nr./dato eller lign.)<br>sesnr. 87207_version 1_2021-11-26 |